CLINICAL TRIAL: NCT04662762
Title: A Nursing Intervention Program Significantly Improves Therapeutic Adherence in Elderly People With Acute Myocardial Infarction: a Randomized Controlled Study
Brief Title: A Nursing Intervention Program to Improve Therapeutic Adherence in Elderly People With Acute Myocardial Infarction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Elena Calvo, Principal investigator, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PR034/16
Record Dates: First submitted 2020-11-28; First posted 2020-12-10 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Medication Adherence; Myocardial Infarction
Keywords: Elderly; Nursing
MeSH Terms: conditions — Medication Adherence; Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: Patients were randomly assigned to a nursing intervention group or a usual care group (1:1).
  Nonprobabilistic, consecutive sampling was carried out with random assignment of the study groups.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The random assignment was made to the "nursing intervention group" and the "usual care group", generating a list using the EPIDAT ® programme. This list contained the patient number and the assignment group. The randomization procedure was performed during hospitalization for AMI. The researcher did not know the assignment list, calling the research unit at the time of each patient inclusion by phone, when they were told to which group they would belong to once the first interview was over.
  The main outcome measured was therapeutic adherence 12 months after admission. This assessment was performed by trained nurses blinded to the group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nursing intervention group (Experimental): An educational interview by trained nurses was performed at three months in patients allocated to the intervention group. The visit was carried out at the hospital. Family and caregivers were also asked to attend this visit for instruction. For patients unable to move, the nursing team went to their home to perform the intervention, or it was conducted by phone. The duration of this interview was approximately 40 minutes and was focused on some measures and recommendations to improve or maintain adherence. Then, there is a reminder call at 6 months.
  Interventions: Other: Nursing intervention programme
- Usual care group (No Intervention): The patient is followed up and regular visits

INTERVENTIONS:
Other: Nursing intervention programme — educational information
  Arms: nursing intervention group

SUMMARY:
The objective of this study was to assess the impact of a nursing intervention on therapeutic adherence in elderly patients after acute myocardial infarction compared to a control group

DETAILED DESCRIPTION:
A comprehensive geriatric assessment was performed during the first admission in all patients. Patients were randomly allocated to a nursing intervention group or a usual care group. In patients from the intervention group, a nursing intervention programme was performed 3 months after admission, based on education, support and patient monitoring to improve therapeutic adherence and a 6 month phone call. The main outcome measured was therapeutic adherence at 12 months, as defined by a combination of adherence measurement tools (Morisky-Green and Hayness-Sacket scales, attendance at visits and withdrawal of medication from the pharmacy). Therapeutic adherence was assessed by nurses blinded to the assignment group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with STEMI aged 75 years or older underwent primary percutaneous coronary intervention (PCI)

Exclusion Criteria:

* Patients who refused to participate in the study
* Patients unable to perform geriatric assessment.
* Patients admitted to nursing homes or social health centres.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 160 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-05-28 (Actual)

PRIMARY OUTCOMES:
Number of patients with therapeutic adherence | 12 months after admission
  The main outcome measured was therapeutic adherence 12 months after admission. The definition of adherence was a single measure taking into account 4 different methods (see below). Patients were considered adherent when the 4 criteria were present (called "global adherence").Measurement unit was: Number of patients with therapeutic adherence
  * Morisky-Green Scale (MGLS): consists of a series of four questions with dichotomous answers (yes/no) that affect the patient's behaviour regarding compliance.
  * Self-reported compliance communication: Haynes-Sackett method: involves asking the patient one question. If the answer is affirmative, is considered adherent.
  * Records of dispensations in the pharmacy: Patients who withdrew all medications during the year were considered adherent.
  * Attendance at scheduled appointments: It is recorded if the patient has missed any of the control visits by both the doctor and the nurse during the first year.

SECONDARY OUTCOMES:
Rate of readmission, | During the 12 months after the admission
  Need for hospital readmission
Rate of visits to the emergency room | During the 12 months after the admission
  Need for emergency visits at hospital
Rate of mortality | During the 12 months after the admission
  Deaths of cardiac origin were those caused by myocardial infarction, sudden death or heart failure.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Calvo, RN, Principal Investigator — Nurse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Calvo E, Izquierdo S, Castillo R, Cesar E, Domene G, Gomez AB, Guerrero C, Andreu-Periz L, Gomez-Hospital JA, Ariza-Sole A. Can an individualized adherence education program delivered by nurses improve therapeutic adherence in elderly people with acute myocardial infarction?: A randomized controlled study. Int J Nurs Stud. 2021 Aug;120:103975. doi: 10.1016/j.ijnurstu.2021.103975. Epub 2021 May 10. PMID 34102371